CLINICAL TRIAL: NCT01088178
Title: Levonorgestrel-Intrauterine System (LNG-IUS) Insertion in the Postpartum Period: A Prospective, Randomized Pilot Study of Three Time Intervals
Brief Title: Levonorgestrel-Intrauterine System (LNG-IUS) Insertion in the Postpartum Period
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No recruitment occurred and the PI stopped the study
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMCP.2009.0062
Record Dates: First submitted 2010-02-25; First posted 2010-03-17 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Contraception
Keywords: Long-Acting Reversible Contraception; Contraceptive Agents; Therapeutic Uses; Contraceptive Agents, Female; Reproductive Control Agents; Pharmacologic Actions; Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Immediate Postplacental (Experimental): Within 10 minutes from delivery of placenta
  Interventions: Device: Levonorgestrel Intrauterine System (LNG-IUS: Mirena, Bayer)
- Early Postpartum (Experimental): After 10 minutes from delivery of placenta but within 48hrs from delivery
  Interventions: Device: Levonorgestrel Intrauterine System (LNG-IUS: Mirena, Bayer)
- Interval (Experimental): After 6 weeks postpartum
  Interventions: Device: Levonorgestrel Intrauterine System (LNG-IUS: Mirena, Bayer)

INTERVENTIONS:
Device: Levonorgestrel Intrauterine System (LNG-IUS: Mirena, Bayer) — Placement of Mirena at given intervals during the postpartum period

SUMMARY:
The investigators study is a prospective randomized trial of women undergoing the levonorgestrel intrauterine system (LNG-IUS: Mirena©, Bayer) at three separate time periods: immediate post placental (IPP) defined as insertion within 10 min delivery of placenta, early post partum (EP) defined as insertion after 10 min but within 72hrs postpartum, or interval (INT) insertion defined as insertion after 6wks postpartum. This is a pilot study in preparation for a multicenter, prospective randomized study of long-acting reversible contraception in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* All reproductive age women who express a desire for the LNG-IUS (Mirena©) at routine questioning at their 36-38 week prenatal appointment or upon admission to labor and delivery are eligible for our study.

Exclusion Criteria:

* Contraindications to the LNG-IUS include: Pregnancy or suspicion of pregnancy, Congenital or acquired uterine anomaly including fibroids if they distort the uterine cavity, Postpartum endometritis within the past 3 months, Known or suspected uterine or cervical neoplasia or unresolved, abnormal pap smear, untreated acute cervicitis or vaginitis including bacterial vaginosis or other lower genital tract infections, acute liver disease or liver tumor, hypersensitivity to any component of the product, known or suspected carcinoma of the breast. Any of these conditions would exclude the patient from our study.
* Delivery <36 weeks
* Intrapartum chorioamnionitis (defined as maternal fever >100.4 and two of the following conditions: Maternal leukocytosis (greater than 15,000 cells/cubic millimeter), Maternal tachycardia (greater than 100 beats/minute), Fetal tachycardia (greater than 160 beats/minute), Uterine tenderness, Foul odor of the amniotic fluid
* Postpartum Hemorrhage (defined as >500cc EBL for spontaneous vaginal delivery)
* Cesarean delivery if randomized to IPP or EP placement

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Continuation Rates of the LNG-IUS when placed postpartum at three time periods | at 6 months
  Determine if there is a difference in continuation rates at 6 months between participants who had the LNG-IUS placed at three different time periods: Immediate Postplacental (within 10 minutes from delivery of placenta), Early Postpartum (after 10 minutes but before 48 hours postpartum) , and Interval (after 6 weeks postpartum).

SECONDARY OUTCOMES:
Expulsion rate of the LNG-IUS when placed postpartum at three time periods | at 3 weeks
  Determine if there is a difference in expulsion rates at the three different time periods of placement.
Pain at placement | at 1 minute
  Determine if there is a difference pain as assessed with the Visual Analog Scale at the time of placement of the LNG-IUS at three time period: Immediate Postplacental, Early Postpartum, or Interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center, Portsmouth, Virginia, United States

REFERENCES:
- [Derived] Dahlke JD, Terpstra ER, Ramseyer AM, Busch JM, Rieg T, Magann EF. Postpartum insertion of levonorgestrel--intrauterine system at three time periods: a prospective randomized pilot study. Contraception. 2011 Sep;84(3):244-8. doi: 10.1016/j.contraception.2011.01.007. Epub 2011 Feb 24. PMID 21843688